CLINICAL TRIAL: NCT05362240
Title: Functional Outcomes of Three Corner Fusion Without Triquetrum Excision Versus Conventional Four Corner Fusion in Scaphoid Non Union Advanced Collapse (SNAC) Wrist Grade II and III : a Prospective Randomized Controlled Trial
Brief Title: Outcomes of Three Corner Fusion Without Triquetrum Excision Versus Conventional Four Corner Fusion in SNAC Wrist
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASU M D 296/2019
Record Dates: First submitted 2022-05-02; First posted 2022-05-05 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Scaphoid Fracture
Keywords: SNAC wrist; Four-corner fusion; Three corner fusion

STUDY DESIGN:
Intervention Model Description: Two groups with the first intervention four corner fusion , and the second with three corner fusion without triquetrum excision
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Four corner fusion (Experimental): Scaphoid excision and fusion between lunate , capitate , hamate and triquetrum using k.wires
  Interventions: Procedure: Four corner fusion
- Three corner fusion without triquetrum excision (Experimental): Scaphoid excision with fusion between lunate , capitate and hamate with preservation of triquetrum
  Interventions: Procedure: three corner fusion without triquetrum excision

INTERVENTIONS:
Procedure: Four corner fusion — First , we inspected the radiocarpal joint for any arthritis before starting the technique , if there was no arthritis , we go on for the procedure . After scaphoid excision , we denuded the articulating surfaces between lunate , capitate , hamate and triquetrum . Then ,any lunate extension deformity was corrected . Then we use k.wires as a fixation method between the above mentioned carpal bones
  Other Names: four corner arthrodesis
  Arms: Four corner fusion
Procedure: three corner fusion without triquetrum excision — First , we inspected the radiocarpal joint for any arthritis before starting the technique , if there was no arthritis , we go on for the procedure . After scaphoid excision , we denude the articulating surfaces between lunate , capitate , hamate and don not include triquetrum. Then ,any lunate extension deformity was corrected . Then we use k.wires as a fixation method between the above mentioned carpal bones.
  Arms: Three corner fusion without triquetrum excision

SUMMARY:
The investigator compare two types of limited wrist arthrodesis used for management of cases with scaphoid non union advanced collapse (SNAC) as regard the outcome to provide the most suitable technique

DETAILED DESCRIPTION:
There is a controversy regarding the suitable limited wrist arthrodesis technique for SNAC wrist grade II and III . For several decades , scaphoid excision and four corner fusion (between lunate , capitate , hamate and triquetrum) was the gold standard with good functional outcomes . Later on , a more limited fusion technique was described , three corner fusion ( between lunate , capitate and hamate) with scaphoid and triquetrum excision to improve ulnar deviation range . On the other hand , biomechanical studies mentioned that the triquetrum had a certain proprioceptive function that could be affected when it was included in the fusion process .Furthermore , if the triquetrum was excised the radiolunate contact pressure would increase with higher risk of development of arthritis. The aim of the study to compare the conventional four corner fusion with three corner fusion with triquetrum excision

ELIGIBILITY:
Inclusion Criteria:

* SNAC wrist G II , III

Exclusion Criteria:

* cases with radiolunate arthritis
* Scapholunate advanced collapse
* Grade 1 Scaphoid non union advanced collapse
* Kienbock disease
* Skeletally immature patients

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-12-02 (Actual)

PRIMARY OUTCOMES:
Range of motion | preoperative
  measuring range of motion and sagittal and coronal plane using goniometer
Range of motion | one year postoperative
  measuring range of motion and sagittal and coronal plane using goniometer
Power grip | preoperative
  Using dynamometer , take the average of three successive measures for injured side and normal side . The grip strength recorded as number between 1-30 (per square inch ) and as a percentage to the contralateral side
Power grip | one year postoperative
  Using dynamometer , take the average of three successive measures for injured side and normal side . The grip strength recorded as number between 1-30 (per square inch ) and as a percentage to the contralateral side

SECONDARY OUTCOMES:
operative time | Intraoperative
  measuring the operative time
Visual analogue scale | preoperative
  Pain assessment using the scale from 0 to 10 , with 0 no pain , 5 moderate pain , 10 worst possible pain
Visual analogue scale | one year postoperative
  Pain assessment using the scale from 0 to 10 , with 0 no pain , 5 moderate pain , 10 worst possible pain .
Patient satisfaction | preoperative
  Modified Mayo wrist score which involves both patient and physician participation. The scale runs from 0 to 100, with 0 representing a worse wrist condition and 100 suggesting a better wrist condition. It assess discomfort, active flexion/extension arc (in contrast to the contralateral side), grip strength (in comparison to the contralateral side), and the capacity to return to regular job or activities.
Patient satisfaction | one year postoperative
  Modified Mayo wrist score which involves both patient and physician participation. The scale runs from 0 to 100, with 0 representing a worse wrist condition and 100 suggesting a better wrist condition. It assess discomfort, active flexion/extension arc (in contrast to the contralateral side), grip strength (in comparison to the contralateral side), and the capacity to return to regular job or activities.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed M Elmahy, Professor, Study Chair — Ain Shams University
Locations (1):
- Ain Shams University , Faculty of medicine, Al ‘Abbāsīyah, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bain GI, Sood A, Ashwood N, Turner PC, Fogg QA. Effect of scaphoid and triquetrum excision after limited stabilisation on cadaver wrist movement. J Hand Surg Eur Vol. 2009 Oct;34(5):614-7. doi: 10.1177/1753193408094923. Epub 2009 Jul 10. PMID 19592604
- [Background] Scobercea RG, Budoff JE, Hipp JA. Biomechanical effect of triquetral and scaphoid excision on simulated midcarpal arthrodesis in cadavers. J Hand Surg Am. 2009 Mar;34(3):381-6. doi: 10.1016/j.jhsa.2008.11.027. PMID 19258133
- [Background] Delattre O, Goulon G, Vogels J, Wavreille G, Lasnier A. Three-Corner Arthrodesis With Scaphoid and Triquetrum Excision for Wrist Arthritis. J Hand Surg Am. 2015 Nov;40(11):2176-82. doi: 10.1016/j.jhsa.2015.07.032. Epub 2015 Sep 26. PMID 26409577